CLINICAL TRIAL: NCT02527252
Title: Benefits of Craniosacral Therapy in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Craniosacral Therapy in Patients With Chronic Low Back Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Dr, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAL-472
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Low Back Pain; Musculoskeletal Manipulations
Keywords: Massage; Craniosacral; Disability Evaluation; Randomized Controlled Trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Craniosacral therapy (Experimental): All treatments were applied by two experienced therapists with a 10-year certification in manipulative therapy after completion of their physical therapy degree and more than 20 years of clinical experience with patients. All patients received the intervention on the day of their initial examination. The techniques took 50 minutes and were conducted as follows:
  * Pelvic Diaphragm Release.
  * Respiratory Diaphragm Release.
  * Thoracic Inlet Release.
  * Hyoid release.
  * Sacral technique for stabilize L5/sacrum.
  * CV-4 Still Point Induction.
  Interventions: Other: Craniosacral therapy
- Classic Massage (Active Comparator): Classics massage protocol was compounded by the following techniques of soft tissues massage: effleurage, petrissage, friction, and kneading. The techniques took thirty minutes.
  Interventions: Other: Classic Massage

INTERVENTIONS:
Other: Craniosacral therapy
  Arms: Craniosacral therapy
Other: Classic Massage
  Arms: Classic Massage

SUMMARY:
The purpose of the current randomized clinical trial was to analyze the effectiveness of craniosacral therapy on disability, pain intensity, kinesiophobia, quality of life, isometric endurance of trunk flexor muscles, mobility, and oxygen saturation, blood pressure, cardiac index, and biochemical estimation of interstitial fluid in individuals with chronic low back pain.

DETAILED DESCRIPTION:
Objective: To analyze the effects of craniosacral therapy on disability, pain intensity, quality of life, and mobility in patients with chronic low back pain.

Design: A single blinded randomized controlled trial. Setting: Clinical setting. Subjects: Sixty-four patients (42 females) with chronic low back pain. Interventions: Patients were randomly assigned to an experimental group (craniosacral therapy group) or a control group (classic massage group).

Main measures: Self-reported disability (Roland Morris Disability Questionnaire - primary outcome; and Oswestry Disability Index), pain intensity (a 10-point Numerical Pain Rating Scale), scale of kinesiophobia (Tampa Scale of Kinesiophobia), isometric endurance of trunk flexor muscles (McQuade Test), lumbar mobility in flexion, and oxygen saturation, blood pressure, cardiac index, and biochemical estimation of interstitial fluid.

ELIGIBILITY:
Inclusion Criteria:

1. LBP for/over three months.
2. age between 18 and 65 years.
3. score equal or superior of four points on the Roland Morris Disability Questionnaire.
4. not currently receiving physical therapy.

Exclusion Criteria:

1. presence of lumbar stenosis
2. diagnosis of spondylolisthesis
3. diagnosis of fibromyalgia
4. treatment with corticosteroid or oral medication within the past two weeks
5. a history of spinal surgery
6. disease of the central or peripheral nervous system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Disability Questionnaire (RMQ) | Changes in 10 weeks and 14 weeks
  It is one of the most used questionnaires for assessing disability due to LBP. This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to LBP including walking, bending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Index (ODI). | 10 weeks and 14 weeks
  The ODI has 10 items referring to activities of daily living that might be disrupted by LBP. Each item is answered on a 6-point Likert scale ranging from "no problem at all" [0] to "not possible" [5]. The total score ranges from 0 to 50.
10-point Numerical Pain Rating Scale | 10 weeks and 14 weeks
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) was used to assess the patients' current level of pain, and the worst and lowest level of pain experienced in the preceding 24 hours.
Tampa Scale of Kinesiophobia (TSK) | 10 weeks and 14 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17-item questionnaire developed to measure the fear of movement and (re)injury.
Isometric endurance of trunk flexor muscles | 10 weeks and 14 weeks
  To test isometric endurance of trunk flexor muscles we used the McQuade test. Subjects were supine with their arms crossed over the chest, hands on the opposite shoulders, hips bent, and knees and feet apart. They were asked to nod and continue to lift their head and shoulders until the inferior angle of the scapula lifted from the table and maintain the position as long as possible.
Lumbar mobility in flexion | 10 weeks and 14 weeks
  Lumbar mobility in flexion was determined by measuring the finger-to-floor distance with a tape.
Hemoglobin Oxygen Saturation | 10 weeks and 14 weeks
  This outcome measure will be assess with Electro Intersticial Scanner
Systolic Blood Pressure | 10 weeks and 14 weeks
  This outcome measure will be assess with Electro Intersticial Scanner
Diastolic Blood Pressure | 10 weeks and 14 weeks
  This outcome measure will be assess with Electro Intersticial Scanner
Hemodynamic (Cardiac Index) | 10 weeks and 14 weeks
  This outcome measure will be assess with Electro Intersticial Scanner
Insterticial Liquid Biochemical Estimation | 10 weeks and 14 weeks
  This outcome measure will be assess with Electro Intersticial Scanner

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almeria, Almería, Almería, Spain

REFERENCES:
- [Result] Green C, Martin CW, Bassett K, Kazanjian A. A systematic review of craniosacral therapy: biological plausibility, assessment reliability and clinical effectiveness. Complement Ther Med. 1999 Dec;7(4):201-7. doi: 10.1016/s0965-2299(99)80002-8. PMID 10709302
- [Result] Downey PA, Barbano T, Kapur-Wadhwa R, Sciote JJ, Siegel MI, Mooney MP. Craniosacral therapy: the effects of cranial manipulation on intracranial pressure and cranial bone movement. J Orthop Sports Phys Ther. 2006 Nov;36(11):845-53. doi: 10.2519/jospt.2006.36.11.845. PMID 17154138
- [Result] Sutherland WG. The cranial bowl. 1944. J Am Osteopath Assoc. 2000 Sep;100(9):568-73. No abstract available. PMID 11057075
- [Result] Castro-Sanchez AM, Mataran-Penarrocha GA, Sanchez-Labraca N, Quesada-Rubio JM, Granero-Molina J, Moreno-Lorenzo C. A randomized controlled trial investigating the effects of craniosacral therapy on pain and heart rate variability in fibromyalgia patients. Clin Rehabil. 2011 Jan;25(1):25-35. doi: 10.1177/0269215510375909. Epub 2010 Aug 11. PMID 20702514
- [Result] Mataran-Penarrocha GA, Castro-Sanchez AM, Garcia GC, Moreno-Lorenzo C, Carreno TP, Zafra MD. Influence of craniosacral therapy on anxiety, depression and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:178769. doi: 10.1093/ecam/nep125. Epub 2011 Jun 15. PMID 19729492
- [Result] Blood SD. The craniosacral mechanism and the temporomandibular joint. J Am Osteopath Assoc. 1986 Aug;86(8):512-9. No abstract available. PMID 3759521
- [Result] Arnadottir TS, Sigurdardottir AK. Is craniosacral therapy effective for migraine? Tested with HIT-6 Questionnaire. Complement Ther Clin Pract. 2013 Feb;19(1):11-4. doi: 10.1016/j.ctcp.2012.09.003. Epub 2012 Nov 9. PMID 23337558
- [Result] Nourbakhsh MR, Fearon FJ. The effect of oscillating-energy manual therapy on lateral epicondylitis: a randomized, placebo-control, double-blinded study. J Hand Ther. 2008 Jan-Mar;21(1):4-13; quiz 14. doi: 10.1197/j.jht.2007.09.005. PMID 18215746
- [Result] Gerdner LA, Hart LK, Zimmerman MB. Craniosacral still point technique: exploring its effects in individuals with dementia. J Gerontol Nurs. 2008 Mar;34(3):36-45. doi: 10.3928/00989134-20080301-04. PMID 18350746